CLINICAL TRIAL: NCT01875315
Title: EXACT-COST: Exercise CMR's Accuracy for Cardiovascular Stress Testing-Comparative Effectiveness of Stress Tests
Brief Title: Comparative Effectiveness of Stress Tests
Acronym: EXACT-COST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Karolina Zareba, MD, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011H0295
Record Dates: First submitted 2013-06-05; First posted 2013-06-11 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Diagnostic Cardiac Imaging

SUMMARY:
The primary objective of this project is to demonstrate that a new approach to cardiac stress imaging that combines treadmill exercise with cardiac magnetic resonance (CMR) provides valuable clinical information in a cost-effective manner.

ELIGIBILITY:
Inclusion Criteria:

* any patient referred for stress SPECT
* known or suspected ischemic heart disease
* ability to perform adequate treadmill stress

Exclusion Criteria:

* any contraindication to MRI (e.g. ferromagnetic foreign body, cerebral aneurysm clip, pacemaker/ICD, severe claustrophobia)
* renal insufficiency (GFR < 40)
* known allergy to gadolinium-based contrast or iodinated contrast (because of the research CTA in patients not referred for cath after 2 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Total patient direct and indirect medical costs for one year following stress testing will be less for patients undergoing stress CMR as compared to patients undergoing stress Nuclear. | baseline
  Patients will undergo either Stress CMR or stress Nuclear testing. For each individual patient, the cost of the initial test, the subsequent follow-up costs, and the total costs over the follow-up period will be calculated. Total costs will be collected for direct medical, direct non-medical and indirect costs. Direct medical costs will include those applied for medications, imaging, invasive therapies and healthcare services; as well as costs resulting from side effects or complications from each of the testing strategies. Direct non-medical costs will include those incurred due to CAD-related illness or the need to seek care, such as caregiver costs and patient transportation costs. Indirect costs, will be defined as lost productivity due to time lost from work, early death or disability.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Dickerson, MD, Principal Investigator — Ohio State University
Locations (4):
- United States (4):
  - Brigham And Womens Hospital, Boston, Massachusetts
  - The Lindner Center at the Christ Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Raman SV, Richards DR, Jekic M, Dickerson JA, Kander NH, Foster EL, Simonetti OP. Treadmill stress cardiac magnetic resonance imaging: first in vivo demonstration of exercise-induced apical ballooning. J Am Coll Cardiol. 2008 Dec 2;52(23):1884. doi: 10.1016/j.jacc.2008.08.046. No abstract available. PMID 19038687
- [Background] Jekic M, Foster EL, Ballinger MR, Raman SV, Simonetti OP. Cardiac function and myocardial perfusion immediately following maximal treadmill exercise inside the MRI room. J Cardiovasc Magn Reson. 2008 Jan 15;10(1):3. doi: 10.1186/1532-429X-10-3. PMID 18272005
- [Background] Foster EL, Arnold JW, Jekic M, Bender JA, Balasubramanian V, Thavendiranathan P, Dickerson JA, Raman SV, Simonetti OP. MR-compatible treadmill for exercise stress cardiac magnetic resonance imaging. Magn Reson Med. 2012 Mar;67(3):880-9. doi: 10.1002/mrm.23059. Epub 2011 Aug 16. PMID 22190228
- [Background] Raman SV, Dickerson JA, Jekic M, Foster EL, Pennell ML, McCarthy B, Simonetti OP. Real-time cine and myocardial perfusion with treadmill exercise stress cardiovascular magnetic resonance in patients referred for stress SPECT. J Cardiovasc Magn Reson. 2010 Jul 12;12(1):41. doi: 10.1186/1532-429X-12-41. PMID 20624294